CLINICAL TRIAL: NCT06752837
Title: Comparing the Efficacy of a Stainless-Steel Rotary File with Two Nickel-Titanium Systems on Periapical Lesion Healing Using Cone-Beam Computed Tomography
Brief Title: Comparing Efficacy of a Stainless-steel Rotary File with Two Nickel-titanium Systems on Periapical Lesion Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beirut Arab University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-H-0056-D-P-0457
Record Dates: First submitted 2024-12-16; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2017-12

CONDITIONS: Periapical Diseases; Root Canal Infection
Keywords: CBCT; Nickel-titanium files; Tornado rotary system
MeSH Terms: conditions — Periapical Diseases | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- The instrumentation was done using a revolving SS Tornado rotary system (MIB, FRANCE). (Experimental): Root canal treatment was done using Stainless steel tornado rotary system
  Interventions: Device: Tornado rotary system; Device: Cone beam computed tomography
- Instrumentation was done using a reciprocating Ni-Ti WaveOne system (Dentsply Maillefer, Ballaigues, (Experimental): Root canal treatment was done using WaveOne rotary system
  Interventions: Device: WaveOne rotary system; Device: Cone beam computed tomography
- The instrumentation was done using a rotative Ni-Ti OneShape system (Micro Mége, Besançon, France). (Experimental): Root canal treatment was done using OneShape rotary system
  Interventions: Device: OneShape rotary system; Device: Cone beam computed tomography

INTERVENTIONS:
Device: Tornado rotary system — In arm one, stainless steel tornado files works by high-speed rotation that influences the fluid dynamics within the canal and improves irrigation efficiency. Canals are finished with a file having a 4% taper and an apical diameter of 0.25 mm.
  Other Names: Revolving SS Tornado rotary system (MIB, FRANCE) in arm one
  Arms: The instrumentation was done using a revolving SS Tornado rotary system (MIB, FRANCE).
Device: WaveOne rotary system — In arm two, WaveOne system is a single reciprocating file system with a heat-treated NiTi Memory Wire (M Wire).It has a taper of 0.08 in apical 3 mm, with a tip diameter of 0.25 mm. in a torque control endodontic handpiece (X smart plus with reciprocation mode)
  Other Names: In arm two, WaveOne single reciprocating file system
  Arms: Instrumentation was done using a reciprocating Ni-Ti WaveOne system (Dentsply Maillefer, Ballaigues,
Device: OneShape rotary system — In arm three, OneShape system utilizes a conventional, continuous rotational motion. It has asymmetric cross-sectional geometry, and traveling waves of motion that are produced along the file's active region. It has a single constant taper of 0.06 and a tip size of 25 with distinct cross-sectional designs along the whole length of the working parts
  Other Names: In arm three, OneShape rotary system
  Arms: The instrumentation was done using a rotative Ni-Ti OneShape system (Micro Mége, Besançon, France).
Device: Cone beam computed tomography — A post-operative CBCT image was obtained and compared to the pre-operative one to assess the impact of canal preparation of each file on the periapical lesion.
  Other Names: Operating teeth were scanned with an axial slice thickness of 0.1 mm using a CBCT (Kodak 9000C) with an 80 kV, 4 mA, 51 × 51 mm field of view, and 0.1/voxel (mm) size.

SUMMARY:
Background: This study used cone-beam computed tomography (CBCT) to compare a stainless-steel Tornado file system with OneShape and WaveOne rotary systems for biomechanical canal preparation as indicated by the healing of periapical lesions.

Methods: Lower molars with necrotic pulps and periapical lesions were arbitrarily divided into three groups (n=20) rendering to three rotary file systems. After root canal treatment, clinical and radiographic assessment of the apical radiolucency was evaluated at one year using pre- and post-instrumentation CBCT images. Statistical analysis was performed to compare the three systems at a p-value of 0.05.

DETAILED DESCRIPTION:
A sample size of 60 subjects (38 females and 22 males) was randomly selected for this randomized clinical research based on a power of 80%, and a significance level of 0.05. The patients should have lower molars with two separate mesial canals, distinct apical foramen, mature apices, and neither cracks nor resorption. Canal curvature for mesial canals ranged from 15° to 45°. The study excluded patients younger than 16 or older than 65, who had diabetes, immune-compromising conditions, or had previous dental work on the working tooth. We informed the patients about the potential risks, discomfort, and potential benefits. Patients who met the inclusion criteria signed a consent form. Table 1 shows the demographics of the study samples. Every patient was evaluated and reviewed through appropriate history taking, clinical examinations, and pre-operative digital radiography. The past dental and medical history, major complaints, and demographic data were recorded. Operating teeth were scanned with an axial slice thickness of 0.1 mm using a CBCT (Kodak 9000C) with an 80 kV, 4 mA, 51 × 51 mm field of view, and 0.1/voxel (mm) size. The patients were then divided randomly into three equal groups (n = 20). After proper anesthesia and isolation, access cavities were completed with a round bur, followed by an Endo Z bur. Working length was determined using an apex locator (DENTA PORT ZX, Japan), and confirmed by periapical X-ray. Canal patency was established with a #15 K-type file (MANI, Vietnam) and RC prep glide path (Premier Dental, USA). Canals were prepared with the assigned instrumentation system according to the manufacturer's instructions and irrigated with 2 mm of a 2.5% sodium hypochlorite solution (NaOCl) (Clorox, Lebanon) followed by 3.0 mL of 17% ethylene-diamine-tetraacetic acid (EDTA) (NEXABIO, Korea) for 1 minute, and then 1.3% NaOCl as final irrigation. Tornado Finisher was used as directed by the manufacturer at 1 mm short of the working length in an up-and-down motion. In the other two groups, irrigation was performed with a 31G side-vented needle (Ultradent Products Inc.) placed passively into the canal, 1 mm short of the working length.Intracanal calcium hydroxide was added to the canals for one week. Every tooth in the three groups underwent the same obturation procedure (Lateral condensation technique) using gutta-percha (DiaDent, Korea) and sealer (META BIOMED, Korea). Finally, coronal preparation of all teeth was restored with composite filling (Ivoclar, Switzerland). Clinical evaluation was conducted at a one-year follow-up visit for each patient including spontaneous pain, sinus tract, swelling, mobility, periodontal probing depths greater than baseline, or sensitivity to percussion or palpation. A post-operative CBCT image was obtained and compared to the pre-operative one to assess the impact of canal preparation of each file on the periapical lesion based on Estrela et al.CBCT periapical index (CBCT PAI). The radiolucent area of the periapical lesion was measured in three dimensions on the CBCT scan. Bucco-palatal, mesiodistal, and diagonal measurements were obtained, and the greatest diameter was recorded for scoring the lesion extension . Measurements were conducted simultaneously and independently by two examiners and any discrepancies were discussed and remeasured for one measurement agreement. Cortical bone expansion (E) and cortical bone destruction (D) were included in the scoring system as appropriate. If either of these conditions was found in the CBCT analysis, the variables E and D were added to each score. Qualitative analysis of clinical evaluations was conducted for signs and symptoms. The pre- and post-operative Estrela et al. index scores were recorded. The Statistical Package for the Social Sciences software (SPSS 22, SPSS Inc, Chicago, IL) was used to perform the statistical analysis. The median was used to describe the qualitative data for all groups and normal distribution was tested using Shapiro-Wilk test. Since the data did not follow a normal distribution, the scores of the size of the apical lesion before and after one year were done for each group using the Wilcoxon signed ranks test while inter-group comparison was done using the Kruskal Wallis test followed by Mann-Whitney test for comparison of pairs. All statistical tests were performed at a p-value of 0.05.

ELIGIBILITY:
Inclusion Criteria:

The patients should have lower molars with

* Two separate mesial canals.
* Distinct apical foramen.
* Mature periapical apices.
* No tooth cracks.
* No root resorption.
* Canal curvature for mesial canals ranged from 15° to 45°.

Exclusion Criteria:

* Patient who is younger than 16 or older than 65.
* Diabetic patient.
* Immune-compromising conditions.
* Patient has previous dental work on the working tooth.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Three-dimension lenght in millimeter for apical radiolucency in CBCT for each pateint | One-year follow-up visit for each pateint
  A post-operative Cone beam computed tomography(CBCT) image was obtained and compared to the pre-operative one to assess the impact of canal preparation of each file on the periapical lesion based on Estrela et al CBCT periapical index (CBCT PAI). The radiolucent area of the periapical lesion was measured in millimeters for the three dimensions on the CBCT scan. Bucco-palatal, mesiodistal, and diagonal measurements were obtained, and the greatest diameter was recorded for scoring the lesion extension. Measurements were conducted simultaneously and independently by two examiners and any discrepancies were discussed and remeasured for one measurement agreement.

SECONDARY OUTCOMES:
Qualitative scoring for clinical criteria for each pateint | One-year follow-up visit for each pateint.
  The scoring description was collected for clinical criteria. The scoring was for the presence or absence of spontaneous pain, sinus tract, swelling, tooth mobility, sensitivity to percussion or palpation and the depth of periodontal probing in millimeter greater than preoperative baseline. Scoring was done for each item using scales according to published previous research in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: alaa eldeen O Mais, PhD, Principal Investigator — Beirut Arab University
Locations (2):
- Lebanon (2):
  - College of dentistry, Beirut Arab University, Beirut
  - faculty of dentistry, Beirut Arab University, Beirut

IPD SHARING:
Plan to Share IPD: No
IPD can't be shared due to ethical issues. IPD of this study is confidential.

REFERENCES:
- [Background] Dorasani G, Madhusudhana K, Chinni SK. Clinical and radiographic evaluation of single-visit and multi-visit endodontic treatment of teeth with periapical pathology: An in vivo study. J Conserv Dent. 2013 Nov;16(6):484-8. doi: 10.4103/0972-0707.120933. PMID 24347878
- [Background] De-Deus G, Souza EM, Barino B, Maia J, Zamolyi RQ, Reis C, Kfir A. The self-adjusting file optimizes debridement quality in oval-shaped root canals. J Endod. 2011 May;37(5):701-5. doi: 10.1016/j.joen.2011.02.001. Epub 2011 Mar 23. PMID 21496675
- [Background] Patel S, Brown J, Pimentel T, Kelly RD, Abella F, Durack C. Cone beam computed tomography in Endodontics - a review of the literature. Int Endod J. 2019 Aug;52(8):1138-1152. doi: 10.1111/iej.13115. Epub 2019 Apr 9. PMID 30868610
- [Background] Estrela C, Bueno MR, Azevedo BC, Azevedo JR, Pecora JD. A new periapical index based on cone beam computed tomography. J Endod. 2008 Nov;34(11):1325-1331. doi: 10.1016/j.joen.2008.08.013. Epub 2008 Sep 17. PMID 18928840
- [Background] Moreinos D, Dakar A, Stone NJ, Moshonov J. Evaluation of Time to Fracture and Vertical Forces Applied by a Novel Gentlefile System for Root Canal Preparation in Simulated Root Canals. J Endod. 2016 Mar;42(3):505-8. doi: 10.1016/j.joen.2015.12.023. Epub 2016 Jan 28. PMID 26831050
- [Derived] Mais AO, Abdallah AM, Osman E, Alhadainy HA. Cone-Beam Computed Tomographic Evaluation of Periapical Lesion Healing After Root Canal Preparation with Different File Systems. Bioengineering (Basel). 2025 Nov 19;12(11):1267. doi: 10.3390/bioengineering12111267. PMID 41301223